CLINICAL TRIAL: NCT01699152
Title: Phase 1 Dose-Escalation and Pharmacokinetic Study of TG02 Citrate in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Phase 1 Study of TG02 Citrate in Patients With Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG02-102
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2016-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TG02 citrate (Experimental): TG02 citrate capsules given orally.
  Interventions: Drug: TG02 citrate

INTERVENTIONS:
Drug: TG02 citrate — TG02 citrate capsules
  Other Names: No other names

SUMMARY:
This is a multi-center, open-label, dose escalation study.

DETAILED DESCRIPTION:
The primary objective is to determine the highest dose of TG02 citrate that can be safely given to patients with Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed Chronic Lymphocytic Leukemia Small Lymphocytic Lymphoma.
* Patients must meet one or more of the following indications for treatment:

  1. Progressive disease or marked splenomegaly and/or lymphadenopathy.
  2. Anemia (hemoglobin <11 mg/dL) or thrombocytopenia (platelets<100,000/μL).
  3. Unexplained weight loss exceeding 10% of body weight over the previous 6 months.
  4. CTCAE Grade 2 or 3 fatigue.
  5. Fevers >100.5º F or night sweats for more than 2 weeks without evidence of infection.
  6. Progressive lymphocytosis, with an increase exceeding 50% over a 2 month period or a doubling time of less than 6 months.
  7. Need for cytoreduction prior to allogeneic stem cell transplant.
* Patients must have relapsed or refractory disease after ≥1 prior line of treatment.
* The interval from prior treatment to time of study drug administration should be at least 5 half-lives for cytotoxic and noncytotoxic agents.
* Low-dose corticosteroids (prednisone <20 mg/ day or equivalent dose) are permitted throughout study.
* Clinically significant toxicities from prior chemotherapy must be resolved to Grade ≤ 1.
* Age >18 years.
* ECOG performance status ≤2.
* Life expectancy ≥ 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count >1,000/μL in absence of bone marrow involvement
  * platelets ≥30,000/μL in absence of bone marrow involvement
  * If patient has extensive bone marrow involvement, minimum ANC and platelet levels are not required.
  * total bilirubin ≤1.5 X institutional ULN unless due to Gilbert's syndrome, controlled autoimmune hemolytic anemia or immune thrombocytopenia
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional ULN unless due to disease
  * creatinine <2.0 mg/dL OR creatinine clearance >50 mL/min/1.73 m2
* Negative serum or urine pregnancy test at the time of first dose for WOCBP.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for required assessments.
* Ability to take oral medication.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (CTCAE Grade > 1) due to agents administered more than 3 weeks earlier.
* Patients who have received prior treatment with a CDK inhibitor within 12 months of study enrollment.
* High-dose corticosteroids (prednisone ≥20mg/day or equivalent dose) must be discontinued ≥ 7 days of initiating therapy.
* Patients with known central nervous system involvement.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as TG02 citrate.
* Patients with G6PD deficiency.
* Concurrent severe or uncontrolled medical disease (including but not limited to history of ventricular arrhythmia or symptomatic conduction abnormality within 12 months, ongoing or active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Pregnant and/or breast-feeding women.
* Prior or second malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, or other cancer for which the subject has received curative therapy at least 3 years prior to study entry.
* Known HIV or AIDs.
* QTc interval prolongation >450ms for males and >470 ms for females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  To assess the number of patients with dose-limiting toxicities (DLT) and the dose of TG02 citrate that can be safely given to patients with CLL or SLL.

SECONDARY OUTCOMES:
Adverse Events | 28 days
  The number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: T Parrott, Study Director — Tragara Pharmaceuticals
Locations (5):
- United States (5):
  - GRU, Augusta, Georgia
  - DFCI, Boston, Massachusetts
  - OSU, Columbus, Ohio
  - SCRI, Nashville, Tennessee
  - MDACC, Houston, Texas